CLINICAL TRIAL: NCT01072812
Title: An Open-Label, Two-Stage Study to Evaluate the Pharmacokinetics and Pharmacodynamics of POSIPHEN® in Plasma and CSF After a 10-Day Treatment Period in Subjects With Amnestic Mild Cognitive Impairment
Brief Title: Study of the Pharmacokinetics and Pharmacodynamics of POSIPHEN® in Subjects With Amnestic Mild Cognitive Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision based on funding
Sponsor: Annovis Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QR 12001
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Alzheimer's Disease; Amnestic Mild Cognitive Impairment
Keywords: Alzheimer's; Amnestic Mild Cognitive Impairment; Pharmacokinetics; Pharmacodynamics; Biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posiphen® tartrate capsules (Experimental)
  Interventions: Drug: Posiphen® tartrate capsules

INTERVENTIONS:
Drug: Posiphen® tartrate capsules — Capsules administered (240 mg/day) for 10 days Capsules administered (160 mg/day) for 10 days
  Other Names: Posiphen® Tartrate

SUMMARY:
This trial will determine the pharmacokinetics of Posiphen® in both plasma and CSF after a 10-day treatment period with Posiphen® in subjects with amnestic MCI. The effects of this treatment on biomarkers will also be determined in CSF, whole blood, and plasma or serum as primary pharmacodynamic (PD) objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Males or post-menopausal females aged 55 to 80 years, inclusive.
2. Must have Mild Cognitive Impairment (MCI) (amnestic subtype) according to Petersen's criteria (2004).
3. Mini Mental Status Examination (MMSE) score should be ≥24.
4. Must score below a pre-determined cut-off score on the logical memory II delayed paragraph recall sub-test of the Wechsler Memory Scale Revised (WMS-R).
5. Must have a Clinical Dementia Rating of 0.5 with a memory box score of 0.5 or 1.0.
6. Modified Hachinski score of less than or equal to 4.
7. Hamilton Depression rating scale (HAMD17) score of less than or equal to 12 with a score of 0 on items 1, 2, and 3 (depressed mood, feelings of guilt, and suicidal ideation).
8. No evidence of current suicidal ideation or previous suicide attempt in past 2 years as evaluated in the Columbia Suicidality Checklist.
9. MRI scans within 12 months prior to screening, or per screening MRI, without evidence of infection, infarction, or other focal lesions and without clinical symptoms suggestive of intervening neurological disease.
10. No clinically significant abnormalities in the lumbar spine should be present on a lumbar X-ray that would contraindicate lumbar puncture.
11. Adequate visual and hearing ability (physical ability to perform all the study assessments).
12. Normal B12, folic acid, and thyroid function tests (thyroid stimulating hormone [TSH], free T4, and free T3).
13. Do not require nursing home care.

Exclusion Criteria:

1. Any significant neurologic disease other than amnestic MCI, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
2. Major depression, schizophrenia or another major psychiatric disorder as described in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) within the past 2 years.
3. Psychotic features, agitation, or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.
4. History of alcohol or substance abuse or dependence within the past 2 years.
5. Subjects with any febrile illness within 1 week prior to the CSF collection.
6. Subjects who have history of migraine headaches and any other type of headaches of at least moderate severity more than twice per month.
7. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol or pose potential risk to the subjects.
8. Use of medications prohibited by the study.
9. Any clinically significant laboratory abnormalities.
10. Subjects with infection or inflammation of the skin or skin disease at or in proximity to the lumbar puncture site.
11. History of lumbar spine surgery or chronic low back pain (CLBP).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 10 days
  To determine the pharmacokinetics (PK) of Posiphen® and its metabolites in plasma and CSF after a 10-day treatment period with Posiphen®.
Pharmacodynamics | 10 days
  To assess the effects of a 10-day treatment period with Posiphen® on the levels of amyloid precursor protein (APP), amyloid β protein 40 (Aβ40), amyloid β protein 42 (Aβ42), acetylcholinesterase (AChE), and butyrylcholinesterase (BChE) in plasma and CSF from subjects with amnestic MCI.

SECONDARY OUTCOMES:
Biomarkers | 10 days
  To assess the effects of a 10-day treatment period with Posiphen® on the levels of amino terminal fragment (N-APP), tau (T-tau), phosphorylated tau (P-tau), nerve growth factor (NGF), brain derived neurotrophic factor (BDNF), interleukin 1B (IL1B), S-100B protein (S-100B) in plasma or serum and CSF, and the activities of AChE and BChE in whole blood or plasma and CSF from subjects with amnestic MCI.
Safety | 10 days
  To determine the safety and tolerability of a 10-day treatment period with Posiphen®.

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Leibowitz, MD, Principal Investigator — CEDRA
Locations (1):
- CEDRA Clinical Research, LLC, San Antonio, Texas, United States